CLINICAL TRIAL: NCT01674751
Title: What to Eat for Lunch? A Pilot Study to Improve Healthier Eating at Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Aramark Healthcare (Unknown)
Responsible Party: Principal Investigator, Etienne Phipps, Director Einstein Urban Health, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HN 4262
Record Dates: First submitted 2012-07-30; First posted 2012-08-29 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2012-08

CONDITIONS: Dietary Habits
Keywords: pre-ordering; healthy eating; mindfulness; incentives; employees
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intervention (Experimental): Group begins the 4 week Pre-Ordering Program intervention immediately following a 4-wk baseline period.
  Interventions: Other: Pre-ordering program
- Wait-listed control (Other): Group begins the 4 week Pre-Ordering Program intervention following an 8-wk baseline period.
  Interventions: Other: Pre-ordering program

INTERVENTIONS:
Other: Pre-ordering program — During the 4 week intervention phase, participants use the pre-ordering program, receive a novel, "smart receipt" upon checkout that will detail the caloric and fat content of what they ordered, and receive price discounts for select low calorie and low fat items. The pre-ordering system is designed to provide the opportunity for the individual to see what is available along with nutritional information and to make a selection ahead of time.

SUMMARY:
This pilot study will test the feasibility and potential effectiveness of a novel approach to improve food choices by employees about what to eat for lunch. The intervention involves the testing of an on-line pre-ordering food program with nutritional information linked to a hospital cafeteria. In this study, the investigators use positive reinforcement of feedback and price discounts during the intervention phase, and then withdraw those components in order to assess the potential for changes to be retained after the study is over.

The study draws on principles from the field of behavioral economics and behavioral change. The investigators test the effectiveness of the intervention with 30 employees (study participants) who are overweight or obese. Based on a recent screening of over 5600 Einstein employees, 66% of those screened were identified as either overweight or obese. There are 3 phases to the trial: baseline (P1), 4 week intervention, (P2) and tapering (intervention without reinforcement) (P3). Participants are randomized to one of two groups (intervention and wait-listed controls).

Our primary hypotheses are that:

1. Participants will purchase lunches with fewer calories during the intervention compared to baseline.
2. Participants will purchases lunches with fewer calories in the tapering phase compared to baseline.

Secondary hypotheses include that, compared with baseline, participants will order lunches with less fat. Changes in participant weight based on self selected goals, and in a measure of mindful eating will also be investigated. The investigators expect that participant adherence will be associated with improved outcomes compared to those who are less adherent.

ELIGIBILITY:
Inclusion Criteria:

* Interested in improving their food choices as it relates to healthier eating and weight loss
* Adult employee at large, urban hospital in Philadelphia at which study is being conducted
* Eats at least 4 lunch meals a week at study cafeteria
* BMI greater than or equal to 25.0 (based on standard classification).
* Willingness to allow researchers to collect data about their lunch purchases
* Willingness to "swipe" their employee card for lunch purchases during the study
* Access to a computer at work
* Capable of providing informed consent
* Has a way of being contacted by telephone, email, fax, or receiving a text message

Exclusion Criteria:

* Planning to terminate hospital employment within the next 4 months
* Individuals unable to consent
* Individuals who are not yet adults
* Employees who are pregnant
* Employees with hypertension, dyslipidemia or coronary artery disease whose medical therapy has changed in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total number of calories | Participants are followed for a minimum of 12 weeks and the total calories from their lunchtime meals are recorded daily.
  The average number of calories (Kcal) purchased for lunch.

SECONDARY OUTCOMES:
Total number of calories from fat | Participants are followed for a minimum of 12 weeks and the total calories from fat in their lunchtime meals are recorded daily.
  The average number of calories from fat (g) purchased for lunch.
Participant adherence | Participants are followed for a minimum of 12 weeks
  Participant adherence is measured by the participants' self-report of engagement in the intervention activities, objective measure of using the pre-ordering system to place lunch purchases, objective measure of the purchase of lunch in the study cafeteria, completion of study materials, and participant report of barriers to engagement in the study.
Participant body weight (kg) | Recorded at the time of recruitment into the study and again following the 8 week intervention
  The average percent change in body weight from baseline to end of the intervention.
Hemoglobin A1c (HbA1c) | Measured at the time of recruitment into the study and again following the 8 week intervention
  The average change in participant Hemoglobin A1c (HbA1c, mmol/mol) will be reported in order to assess change in average plasma glucose concentrations.
Cholesterol subfractions | Measured at the time of recruitment into the study and again following the 8 week intervention
  The average change in participant cholesterol subfractions (g/mL) will be reported in order to evaluate change in risk of coronary heart disease.
Blood pressure (mmHg) | Measured at the time of recruitment into the study and again following the 8 week intervention
  The average change in blood pleasure (mmHg) will be reported.
Mindful eating score on 28-item self-report measure | Recorded at the time of recruitment into the study and again following the 8 week intervention
  The average change in mindfulness when eating will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne J Phipps, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States